CLINICAL TRIAL: NCT04276779
Title: Acute Use of Alcohol and Attentional Bias Towards Suicide: An Experimental Test of the Attention-Allocation Model
Brief Title: Effects of Alcohol and Mood on Attention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to the PI leaving the institution. The grant was ended early.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Caitlin Wolford Clevenger, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: GRANT13018273
Record Dates: First submitted 2020-02-14; First posted 2020-02-19 (Actual); Results first posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Suicidal Ideas
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Negative Mood (Experimental)
  Interventions: Other: Alcohol administration; Behavioral: Negative mood induction
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo administration; Behavioral: Negative mood induction
- Positive Mood (Active Comparator)
  Interventions: Other: Alcohol administration; Behavioral: Positive mood induction
- Alcohol (Experimental)
  Interventions: Other: Placebo administration; Behavioral: Positive mood induction

INTERVENTIONS:
Other: Alcohol administration — Participants in the alcoholic beverage group will be provided a dose of 95% alcohol (0.99g/kg for males and 0.90 g/kg for females body weight) distributed in two equally spaced beverages (mixed with orange juice 1:5 ratio). This dose will produce a breath alcohol content ranging between .08-.10.
  Arms: Negative Mood; Positive Mood
Other: Placebo administration — Individuals in the placebo condition will receive orange juice with 4 ml of alcohol layered on top of the juice. Ethanol will be sprayed on the rims of the glasses.
  Arms: Alcohol; Placebo
Behavioral: Positive mood induction — Participants will be randomized to either positive mood induction procedure. Both conditions involve listening to music that reliably induces positive mood, while simultaneously reading self-referent statements that also induce either positive mood. This procedure lasts about 10 minutes and produces a transient mood state that passes by the end of the study.
  Arms: Alcohol; Positive Mood
Behavioral: Negative mood induction — Participants will be randomized to either negative mood induction procedure. Both conditions involve listening to music that reliably induces sad mood, while simultaneously reading self-referent statements that also induce either sad mood. This procedure lasts about 10 minutes and produces a transient mood state that passes by the end of the study.
  Arms: Negative Mood; Placebo

SUMMARY:
Acute use of alcohol is related to increased risk for suicide. However, our understanding of this problem is hindered by the lack of experimental tests of conditions underlying the alcohol use-suicide relationship. The attention allocation model (AAM) proposes that alcohol intoxication limits individuals' focus to salient cues in their environment. Thus, acute use of alcohol (AUA) during negative mood states may cause people to focus their attention towards suicide-related cues in their environment, thus increasing their risk for suicide while intoxicated. The proposed pilot study tests the AAM by exploring the combined effects of AUA, mood, and alcohol expectancies on attentional bias towards suicide-related cues. The proposed study will explore the combined impact of AUA and negative mood on attentional bias towards suicide in a sample of community adults. The investigators will further explore whether individual differences in alcohol expectancies influence these associations. The investigators will conduct a 2 by 2 (alcohol/placebo by negative mood/positive mood), between-subjects experiment involving alcohol administration, a well-established mood induction paradigm, and a performance-based dependent measure of attention towards suicide-related cues. The investigators expect that individuals in the negative mood-alcohol condition to show the greatest suicide-related attentional bias. The investigators expect that alcohol expectancies related to suicide will strengthen this association, and that positive mood alcohol expectancies will weaken this association. This pilot study will provide an initial test of the feasibility of this project and the hypotheses. This study will form the basis for a larger scale study able to test the effects.

DETAILED DESCRIPTION:
This is a pilot study designed to explore the combined effects of acute use of alcohol, mood, and alcohol expectancies on attentional bias towards suicide. Community adults (n = 120) will be recruited from the University of Alabama at Birmingham campus and greater Birmingham area through distribution of flyers and posts to social media sites (i.e., Facebook and Craigslist). The investigators are recruiting individuals who are ages 21-65, generally healthy, without current psychiatric disorders, distress, or suicidal ideation, and able to safely consume alcohol. Interested individuals will telephone our research lab, and an initial telephone screening will take place to exclude ineligible participants. Eligible participants will attend an initial study session (lasting about one hour), where informed consent will be obtained,eligibility criteria will be more thoroughly assessed, and baseline measures (e.g., alcohol expectancies) will be completed. Participants who remain eligible will be scheduled for a second session, lasting between 3-10 hours (depending on condition), and will be randomly assigned (individually) to an alcohol condition (alcohol-placebo) and a mood condition (negative-positive mood). Participants in the alcohol condition will be administered alcoholic beverages that will raise their breath alcohol content to .08. Participants in the placebo condition will be told they are receiving alcohol but will receive a nonalcoholic beverage that smells and tastes like alcohol. Participants will participate in a mood induction procedure that involves listening to music and reading statements about the self that are designed to induce a temporary mood state (positive or negative). Immediately following the mood induction, participants will rate their mood using a rating scale and then will complete a computerized assessment of their attentional bias towards suicide-related words (i.e., the Suicide Stroop). This measure involves naming colors of words that vary in meaning (neutral, happy, depressed, and suicide-related words). Participants' response times to name the color of suicide-related words are compared to response times to name neutral words, creating a score of suicide-related attentional bias. Following completion of this task, individuals in the placebo condition will complete a post-study interview, where their experiences and the effectiveness of deception will be assessed. Participants will be debriefed and the deception and reasons for it will be revealed. Participants' suicide risk will be assessed and they will be allowed to leave if risk is low (which the investigators anticipate will be the case for all participants). Individuals in the alcoholic beverage condition will complete the same post-study procedures but after their breath alcohol content lowers to .03. While awaiting their breath alcohol content to lower, these participants will be provided with a comfortable area to rest and watch or read entertainment. They will be provided a full meal and nonalcoholic beverages and will be encouraged to drink some water. Participants' driver's license or government-issued ID will be held by study personnel until their breath alcohol content lowers to .03. Participants will not be allowed to leave until their breath alcohol content lowers to .03, and they pass a field sobriety test. All participants will be provided with cab fare for a safe ride home. Safety checks will be performed for all participants the evening of, day following, and week following the study appointment.

This study was ended prior to the planned study end date due to PI leaving the insitution. Thus only the results for the preliminary data are reported.

ELIGIBILITY:
Inclusion criteria:

1. be between the ages of 21 and 65
2. have consumed an average of at least five or more (four or more for females) standard alcoholic drinks per occasion once over the past year
3. have self-administered a quantity of alcohol that is equal to or greater than the dose that will be administered in the lab on at least three occasions in the past year
4. be able to read and write in English fluently.

Exclusion criteria:

1. active psychosis, suicidal ideation/intent, or mania; currently receiving psychiatric treatment; have received psychiatric treatment in past year or currently experiencing significant psychiatric distress
2. in treatment or recovery from drug or alcohol use disorders or abstaining from alcohol
3. any suicide attempt history
4. pregnant/breast-feeding or immediate plans to become pregnant
5. any chronic health problems or medications that would preclude the use of alcohol
6. (to minimize adverse reactions to alcohol/inappropriate alcohol dose) < 6 feet tall and over 230 lbs., or > 6 feet tall and over 250 lbs.
7. color-blind or sight-impaired
8. knowing someone who has participated in this study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Caitlin Clevenger, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

RESULTS

PARTICIPANT FLOW:
Groups:
- Alcohol and Negative Mood: Alcohol administration: Participants in the alcoholic beverage group will be provided a dose of 95% alcohol (0.99g/kg for males and 0.90 g/kg for females body weight) distributed in two equally spaced beverages (mixed with orange juice 1:5 ratio). This dose will produce a breath alcohol content ranging between .08-.10.
  Negative mood induction: Participants will be randomized to either negative mood induction procedure. Both conditions involve listening to music that reliably induces sad mood, while simultaneously reading self-referent statements that also induce either sad mood. This procedure lasts about 10 minutes and produces a transient mood state that passes by the end of the study.
- Placebo and Negative Mood: Placebo administration: Individuals in the placebo condition will receive orange juice with 4 ml of alcohol layered on top of the juice. Ethanol will be sprayed on the rims of the glasses.
  Negative mood induction: Participants will be randomized to either negative mood induction procedure. Both conditions involve listening to music that reliably induces sad mood, while simultaneously reading self-referent statements that also induce either sad mood. This procedure lasts about 10 minutes and produces a transient mood state that passes by the end of the study.
- Alcohol and Positive Mood: Alcohol administration: Participants in the alcoholic beverage group will be provided a dose of 95% alcohol (0.99g/kg for males and 0.90 g/kg for females body weight) distributed in two equally spaced beverages (mixed with orange juice 1:5 ratio). This dose will produce a breath alcohol content ranging between .08-.10.
  Positive mood induction: Participants will be randomized to either positive mood induction procedure. Both conditions involve listening to music that reliably induces positive mood, while simultaneously reading self-referent statements that also induce either positive mood. This procedure lasts about 10 minutes and produces a transient mood state that passes by the end of the study.
- Placebo and Positive Mood: Placebo administration: Individuals in the placebo condition will receive orange juice with 4 ml of alcohol layered on top of the juice. Ethanol will be sprayed on the rims of the glasses.
  Positive mood induction: Participants will be randomized to either positive mood induction procedure. Both conditions involve listening to music that reliably induces positive mood, while simultaneously reading self-referent statements that also induce either positive mood. This procedure lasts about 10 minutes and produces a transient mood state that passes by the end of the study.
Period: Overall Study
Arm/Group | Alcohol and Negative Mood | Placebo and Negative Mood | Alcohol and Positive Mood | Placebo and Positive Mood
Started | 6 | 6 | 7 | 7
Completed | 6 | 6 | 7 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcohol and Negative Mood | Placebo and Negative Mood | Alcohol and Positive Mood | Placebo and Positive Mood | Total
Number analyzed (Participants) | 6 | 6 | 7 | 7 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.67 (7.71) | 28.17 (8.50) | 28.50 (9.31) | 39.71 (18.51) | 31.84 (12.51)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: data were missing for one participant.
  Participants
    number analyzed (Participants) | 6 | 6 | 6 | 7 | 25
    Female | 2 | 5 | 4 | 5 | 16
    Male | 4 | 1 | 2 | 2 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — The columns (race/ethnicity counts) may not add up to the number in the condition, as participants were given the option to select more than one race/ethnicity. The categories are not mutually exclusive.
  Participants
    East Asian | 1 | 0 | 0 | 1 | 2
    Black/African American | 1 | 1 | 2 | 2 | 6
    White/European Origin | 4 | 5 | 4 | 4 | 17
    South Asian | 1 | 0 | 0 | 0 | 1
    Unknown | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 7 | 7 | 26
Sexual orientation [Count of Participants; unit: Participants] — Population: Missing data for one participant.
  Participants
    number analyzed (Participants) | 6 | 6 | 6 | 7 | 25
    Asexual | 0 | 0 | 0 | 1 | 1
    Heterosexual | 4 | 6 | 6 | 6 | 22
    Gay | 1 | 0 | 0 | 0 | 1
    Bisexual | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Modified Suicide Stroop Task
Description: A computer-based task that assesses reaction time to naming colors of words presented sequentially. Words are suicide, depressive, positive, and neutral-related. Reaction times that are higher indicate that the content of the word interfered with naming the color (i.e., attentional bias). A score is computed that subtracts reaction time to neutral words from that to suicide words, creating a measure of suicide-related attentional bias.
  Minimum total score within sample: -113.00 Maximum total score within the sample: 145.92
  Higher values indicate more attentional bias (worse outcome).
Time Frame: 10 minutes
Population: randomized participants
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Alcohol and Negative Mood | Placebo and Negative Mood | Alcohol and Positive Mood | Placebo and Positive Mood
Number analyzed (Participants) | 6 | 6 | 7 | 7
milliseconds | -10.04 (81.21) | 20.05 (39.49) | 10.08 (55.22) | 6.78 (71.38)

2. Secondary Outcome: Brief Hopelessness Measure (Brief-H-Neg)
Description: A brief, 2-item questionnaire that assesses state hopelessness will also be assessed. The items were rated on a scale of 1 to 5. The scale score was the sum of the two items. The total possible score for the scale (sum of the two items) ranged from 2 to 10.
  Higher values indicate a worse outcome.
Time Frame: 5 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Alcohol and Negative Mood | Placebo and Negative Mood | Alcohol and Positive Mood | Placebo and Positive Mood
Number analyzed (Participants) | 6 | 6 | 7 | 7
score on a scale | 3.17 (2.40) | 3.33 (1.51) | 2.57 (1.13) | 2.29 (0.76)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the baseline visit to one week post final visit (session 2, experimental session involving mood manipulation and beverage administration, up to one month post-baseline visit).
Arm/Group | Negative Mood | Placebo | Positive Mood | Alcohol
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13 | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/14 | 0/13

LIMITATIONS AND CAVEATS:
Please note that this study was terminated. Data collection ended prematurely due to the PI leaving the institution. Preliminary data are reported on the sample collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT04276779/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT04276779/SAP_001.pdf
  • Informed Consent Form (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/79/NCT04276779/ICF_002.pdf